CLINICAL TRIAL: NCT07305870
Title: Effectiveness of Sequential Compression Device and Range of Motion Exercises on Distributive Peripheral Edema and Hemodynamic Stability Among Patients in Critical Care Units
Brief Title: Sequential Compression Device and Range of Motion Exercises on Distributive Peripheral Edema and Hemodynamic Stability Among Patients in Critical Care Units
Acronym: SCD and ROM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karbala University (Other)
Responsible Party: Principal Investigator, Hussein Hamza Jawad, Masters graduate student, Ministry of Health, Iraq
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: uok.coN.25.099
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Edema

STUDY DESIGN:
Intervention Model Description: Sequential Compression Device (SCD) protocol involves a pump linked to calf and thigh braces with individual tubes, applying moderate pressure of approximately 60mmHg through a graduated air chamber in a sequential cycle across four compartments. The inflation lasts for 12 seconds followed by a 48-second deflation, with sessions lasting 2 hours daily for 5 consecutive days.
  The Range of Motion (ROM) Exercises program entails 20 minutes of flexion-extension movements for both limbs, conducted in two sessions per day over 5 days. Patients perform passive range of motion exercises for upper extremities including movements of fingers, wrists, elbows, and shoulders, as well as for lower extremities encompassing toe, ankle, knee, and hip movements.
  In addition control group will receive slandered care which is limps elevation
Masking Description: non
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential Compression Device group (Active Comparator): Sequential Compression Device (SCD) participants group involves a pump linked to calf and thigh braces with individual tubes, applying moderate pressure of approximately 60mmHg through a graduated air chamber in a sequential cycle across four compartments. The inflation lasts for 12 seconds followed by a 48-second deflation, with sessions lasting 2 hours daily for 5 consecutive days.
  Interventions: Device: Sequential compression device
- Range of Motion exercises (Active Comparator): The Range of Motion (ROM) Exercises program entails 20 minutes of flexion-extension movements for both limbs, conducted in two sessions per day over 5 days. Patients perform passive range of motion exercises for upper extremities including movements of fingers, wrists, elbows, and shoulders, as well as for lower extremities encompassing toe, ankle, knee, and hip movements. In addition control group will receive slandered care which is limps elevation
  Interventions: Device: legs exercises

INTERVENTIONS:
Device: Sequential compression device — Sequential Compression Device (SCD) protocol involves a pump linked to calf and thigh braces with individual tubes, applying moderate pressure of approximately 60mmHg through a graduated air chamber in a sequential cycle across four compartments. The inflation lasts for 12 seconds followed by a 48-second deflation, with sessions lasting 2 hours daily for 5 consecutive days.
  Arms: Sequential Compression Device group
Device: legs exercises — The Range of Motion (ROM) Exercises program entails 20 minutes of flexion-extension movements for both limbs, conducted in two sessions per day over 5 days. Patients perform passive range of motion exercises for upper extremities including movements of fingers, wrists, elbows, and shoulders, as well as for lower extremities encompassing toe, ankle, knee, and hip movements. In addition control group will receive slandered care which is limps elevation
  Arms: Range of Motion exercises

SUMMARY:
Objectives of The Study:

1. Assess the effectiveness of sequential compression device on distributive peripheral edema and hemodynamic stability for patients in critical care units.
2. Assess the effectiveness of range of motion on distributive peripheral edema and hemodynamic stability for patients in critical care units.
3. Evaluate the synergic effectiveness of sequential compression device and range of motion on distributive peripheral edema and hemodynamic stability for patients in critical care units
4. Find out the differences between the effectiveness of sequential compression device, range of motion, and synergic effectiveness of both interventions on distributive peripheral edema and hemodynamic stability
5. Find out relationships between the effectiveness of sequential compression device, range of motion, and synergic effectiveness of both interventions with patients' demographic characteristics.

DETAILED DESCRIPTION:
Globally, approximately (13-20) million people treated in intensive care units (ICUs) each year, where common complications such as edema are due to prolonged immobility and critical illness . Edema refers to accumulation of excess fluid in body tissues, manifesting in multi forms such as cerebral, pulmonary, or ocular edema. Peripheral edema considered one of the most prevalent types, specifically represents to swelling in the limbs. It caused by imbalance between oncotic and hydrostatic pressures, leading to increased capillary permeability and fluid accumulation in the interstitial space(Smith et al., 2024).

A study found that hospital mortality was significantly higher in those presenting with peripheral edema (22.2%) compared with those without (12.6%) among 12,778 critically ill patients. Also, the severity of edema at admission correlated with increased mortality risk.

The prevalence of peripheral lower limb edema among older adults in U.S was 20.0%, 19.4%, 19.0%, 19.0%, and 19.1% in 2000, 2004, 2008, 2012, and 2016, respectively. It was significantly associated with clinical, demographic, and lifestyle factors, including obesity, diabetes, hypertension, pain, low physical activity, mobility limitations, advanced age, female sex, minority race, and low socioeconomic status.

In Japan, the Ministry of Health, Labor, and Welfare reported an increase in the number of patients with severe motion disabilities, particularly among individuals over 60 years old. Similarly, data from the Health and Retirement Study revealed that chronic peripheral edema affects approximately 19% to 20% of older adults, particularly among women, racial minorities, and individuals with limited mobility.

Peripheral edema is a multifactorial and complex condition that affects patients suffering from a various of diseases. Its underlying pathology varies considerably, with common causes including congestive heart failure (CHF), liver disease, vascular conditions such as chronic venous insufficiency, and postoperative surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who were hospitalized in critical care units.
* Subjects over the age of 18 years.
* Presence of peripheral edema (pitting edema ≥1+ in lower extremities).
* Patients how are hemodynamically stable.
* Patients how are able to tolerate positioning for interventions.

Exclusion Criteria:

* Patients with lymphedema.
* Patients with chronic kidney disease.
* patients with presence of deep vein thrombosis, severe peripheral arterial disease, or phlebitis.
* patients with open wounds, ulcers, or skin infections on lower limbs.
* patients with fractures, orthopedic surgery, or joint immobility in lower extremities.
* patients with severe cardiac failure or pulmonary edema.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Peripheral edema | The degree of edema will be measured before applying interventions and after 5 consecutive days if study
  Firstly, the edema of lower extremities was measured for all patients in critical care units through pitting edema scale before selecting the participants, then the patients selected for the current study had pitting edema scale >+1. Also, leg circumference had measured by using tape measurement.
Hemodynamic Stability | Hemodynamic parameters will be measured before applying interventions and after 5 consecutive days if study
  Hemodynamic parameters were also assessed before interventions. The Hemodynamic parameters that include the heart rate, blood pressure, respiratory rate, urine output and saturation of oxygen was measured by observation of the reading on the monitoring device that was used in critical care units and attached to the patient, the reading was documented by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein H Jawad MGS study principal investigator, Principal Investigator — Kerbala health department
Locations (1):
- Kerbala health department, Karbala, Center, Iraq

IPD SHARING:
Plan to Share IPD: No